CLINICAL TRIAL: NCT05730166
Title: Conditioned Pain Modulation Induced by Mechanical Stimulation. A Mechanism of Manual Therapy Analgesia: Study 2
Brief Title: Pain Inhibitory Effects of Other Pain Induced by Mechanical Pressure at Different Intensities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josue Fernandez Carnero (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MechCPM2
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Conditioned Pain Modulation; Manual Therapy; Physiotherapy; Physical therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mechanical stimulation at moderate pain intensity (Experimental): Mechanical compression is applied with the thumb to the upper trapezius muscle on the non-dominant side at the midpoint between the acromion and C7. The intensity of this will be regulated by the pain it causes the patient, trying to ensure that it is at all times approximately 5/10 on the numerical pain rating scale (NPRS) with 0 being "no pain at all" and 10 being "the worst pain imaginable". The stimulation will be carried out for 2 minutes.
  Interventions: Other: Mechanical Conditioning stimulus
- Mechanical stimulation at mild pain intensity (Active Comparator): Mechanical compression is applied with the thumb to the upper trapezius muscle on the non-dominant side at the midpoint between the acromion and C7. The intensity of this will be regulated by the pain it causes the patient, trying to ensure that it is at all times approximately 2/10 on the numerical pain rating scale (NPRS) with 0 being "no pain at all" and 10 being "the worst pain imaginable". The stimulation will be carried out for 2 minutes.
  Interventions: Other: Mechanical Conditioning stimulus
- Painless mechanical stimulation (Active Comparator): Mechanical compression is applied with the thumb to the upper trapezius muscle on the non-dominant side at the midpoint between the acromion and C7. The intensity of this will be regulated by the pain it causes the patient, trying to ensure that it is at all times approximately 0/10 on the numerical pain rating scale (NPRS) with 0 being "no pain at all" and 10 being "the worst pain imaginable". The stimulation will be carried out for 2 minutes.
  Interventions: Other: Mechanical Conditioning stimulus

INTERVENTIONS:
Other: Mechanical Conditioning stimulus — Mechanical stimulus on the upper trapezius of the non-dominant side.

SUMMARY:
The objective is to estimate the effects on pain thresholds of a painful mechanical stimulus on the upper trapezius at moderate intensity compared to mild intensity or non-painful.

DETAILED DESCRIPTION:
The mechanical stimulus produced in manual therapy (MT) techniques elicits neurophysiological responses within the peripheral and central nervous system responsible for pain inhibition. Almost all types of MT elicit a neurophysiological response that is associated with the descending pain modulation circuit. But it has not been demonstrated whether this inhibition occurs through a conditioned pain modulation mechanism induced by painful mechanical stimulation that is carried out with manual therapy techniques.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female between 18 and 65 years
* Free of pain and with no history of chronic pain

Exclusion Criteria:

* Pregnant or having given birth within the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Tibialis Anterior Pressure Pain Threshold (PPT) to immediate post-conditioning stimulus | At baseline and immediately after the conditioning stimulus
  PPTs will be assessed on the dominant side over the tibialis anterior muscle using a digital algometer (Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful.The average of 3 assessments on the tibialis anterior of the dominant side will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández Carnero, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain